CLINICAL TRIAL: NCT06821880
Title: Developing a Patient-Reported Outcome (PRO) Screening Measure for Infections and Measuring Quality of Life in Hematological Patients With Secondary Immunodeficiency (SID) Across the Treatment Trajectory - The PRO SID Project
Acronym: PRO-SID
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: 1179/2024; ISR-2022-200331 (Other Grant/Funding Number: Takeda Pharma Ges.m.b.H and Takeda Pharma Vertrieb GmbH & Co. KG as Investigator Initiated Research)
Record Dates: First submitted 2025-01-23; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Chronic Lymphocytic Leukaemia (CLL); Multiple Myeloma (MM); Secondary Immunodeficiency (SID)
Keywords: Chronic Lymphocytic Leukaemia (CLL); multiple myeloma (MM); Secondary immunodeficiency (SID); Infection-related symptoms; Infections; PRO measure; Patient-reported outcomes
MeSH Terms: conditions — Leukemia, B-Cell; Multiple Myeloma; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with MM or CLL at risk of infectious complications due to SID

SUMMARY:
The goal of this observational study is to improve the treatment of hematological patients with secondary immunodeficiency (SID) by developing a patient-reported outcome (PRO) instrument to detect clinically diagnosed infections. The study focuses on adults diagnosed with chronic lymphocytic leukemia (CLL) or multiple myeloma (MM) who are at increased risk of infections due to SID.

The main questions it aims to answer are:

1. Can a newly developed PRO screening tool for infection-related symptoms reliably detect infections in patients with SID?
2. How does the health-related quality of life change over the treatment course

Participants will:

* Complete daily electronic PRO questionnaires (ePRO) to monitor infection-related symptoms
* Complete ePRO health-related quality of life questionnaires every 1.5 months
* Participate in study visits every three months to ensure documentation of clinical data

DETAILED DESCRIPTION:
The aim of this observational study is to develop an ePRO symptom monitoring tool to identify infections among patients with MM or CLL who recently started an anticancer therapy.

This multicenter trial, conducted in participating sites in Germany in Austria, targets a total of 120 adult patients to complete daily ePRO questions in a mobile app regarding current infection-related symptoms.

Objectives:

Primary:

To develop and evaluate the diagnostic accuracy of a newly developed PRO screening measure for detecting clinically diagnosed infections in hematological patients with SID.

Secondary:

To measure QoL over time using validated instruments such as the EORTC QLQ-C30 and disease-specific modules (QLQ-MY20 for MM and QLQ-CLL17 for CLL).

Explore whether PRO-based infection detection prompts subsequent initiation of immunoglobulin replacement therapy (IgRT) and examine QoL before and after its initiation.

Exploratory Objectives:

* To evaluate the completion and adherence rates for ePRO assessments.
* To investigate the predictive value of the PRO screening tool for infection incidence.

To develop a reliable item list to monitor and detect infections, it is necessary to establish a high-quality measurement of infections as criterion. We developed the item list based on items from the European Organisation for Research and Treatment of Cancer (EORTC) Item Library and in line with international best-practice recommendations for item list development. The development comprised a comprehensive review of the literature and existing measures measuring infection-related symptoms, as well as physician input on which domains and symptoms were the most relevant to assess to monitor for infections in this population.

Clinicians will also document any diagnosed infections and relevant clinical data throughout study visits, which take place every three months. These include updates on treatment regimens, disease staging, and infection history.

The app was developed based on the Computer-based Health Evaluation System (CHES) software platform, which allowed for real-time symptom tracking and data integration. The software has been used extensively and also been tested with patients with hematological diseases in the past. For the PRO-SID app, we developed study-specific content, which comprised information in lay language on the diseases (MM and CLL), information on infections and SID, and information on the study itself. The native app (iOS and Android) prompts patients to complete the item list once daily via push-reminders (up to two reminders).

Usability of the app and understanding of the item list within the daily ePRO assessment on infection symptoms has been assessed within a designed feasibility study according to best practice guidelines (data to be published separately). After completion of the feasibility study, we implemented changes to the app based on patients' feedback and answers in the evaluation questionnaires in order to improve the app for the final study.

Patient Safety and Ethics:

The study is conducted in compliance with the Declaration of Helsinki and Good Clinical Practice standards. Informed consent is obtained, and all participant data is de-identified and securely stored to ensure confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>=18 years of age)
* Access to an internet device (e.g., personal computer or tablet to use a web-based platform, or smartphone where the study app can be installed - all common iOS and Android systems)
* German-speaking
* Diagnosis of multiple myeloma or chronic lymphocytic leukemia
* Secondary immunodeficiency (defined as: recurrent infections, infections requiring inpatient treatment, hypogammaglobulinemia, neutropenia and/or lymphopenia on differential blood cell counts, deficit in lymphocyte subsets as assessed by flow cytometry)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are subjects with MM or CLL and a SID who have recently started a anticancer therapy in Germany and Austria.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the ePRO monitoring instrument for infection-related symptoms | From enrollment until study discontinuation or up until study completion (day 365), which ever occurs first
  Evaluation of diagnostic accuracy of the daily ePRO screening measure to detect infections as diagnosed by a clinician (CTCAE).

SECONDARY OUTCOMES:
Changes in health-related quality of life measured with the EORTC QLQ-C30 | From enrollment until study discontinuation or up until study completion (day 365), which ever occurs first
  Changes in health-related quality of life over the study period (from inclusion to six and 12 months) measured with the EORTC Core Quality of Life questionnaire (EORTC QLQ-C30).
Changes in health-related quality of life measured with the EORTC QLQ-MY20 | From enrollment until study discontinuation or up until study completion (day 365), which ever occurs first
  Changes in health-related quality of life over the study period (from inclusion to six and 12 months) measured with the EORTC disease-specific module QLQ-MY20 - a 20 item instrument designed to assess the quality of life of patients with multiple myeloma.
2. Changes in health-related quality of life measured with the EORTC QLQ-CLL17 | From enrollment until study discontinuation or up until study completion (day 365), which ever occurs first
  Description: Changes in health-related quality of life over the study period (from inclusion to six and 12 months) measured with the EORTC disease-specific module QLQ-CLL17 - a 17 item instrument designed to assess the quality of life of patients with chronic lymphocytic leukemia.

CONTACTS AND LOCATIONS:
Locations (5):
- Austria (3):
  - Medizinische Universität Innsbruck, Innsbruck, Tyrolia
  - Medizinische Universität Graz, Graz
  - BKH Kufstein, Kufstein
- Germany (2):
  - Onkologischer Schwerpunkt am Oskar-Helene-Heim, Berlin
  - Klinikum Garmisch-Partenkirchen, Garmisch-Partenkirchen

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: Beginning with publication and ending 10 years after the publication of results
Access Criteria: Open access available